CLINICAL TRIAL: NCT03696927
Title: Active Powered Prosthesis (APEX) for Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AbiliTech Medical Inc. (Industry)
Collaborators: Allina Health System (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 6100003-100 Rev A; R43HD094440 (NIH)
Record Dates: First submitted 2018-09-17; First posted 2018-10-05 (Actual); Results first posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-10

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- User Focus Group Participants (Experimental): Target user population will be human subjects with spinal cord injury at levels C3 to C5, and ASIA Impairment Scale (AIS) A, B, or C.
  Interventions: Device: Active Powered Prosthesis (APEX) for Spinal Cord Injury

INTERVENTIONS:
Device: Active Powered Prosthesis (APEX) for Spinal Cord Injury — The Active Powered Prosthesis (APEX) is a proof-of-concept shoulder-elbow-wrist device intended to provide non-invasive active powered robotic assistive movement to upper extremities. Focus group participants will control the APEX device on a test manikin and provide feedback on the device design and function.

SUMMARY:
The Active Powered Prosthesis (APEX) (AbiliTech Medical Inc., Minneapolis, MN) is a proof-of-concept shoulder-elbow-wrist device intended to provide non-invasive active powered robotic assistive movement to upper extremities. The objective of this study is to perform focus groups with users and clinicians to evaluate a proof of concept active powered assistance device.

ELIGIBILITY:
Inclusion Criteria:

1. Spinal cord injury at levels C3 to C5, and AIS A, B, or C
2. Greater than 3-months post injury or surgery to the spinal column, arms, or shoulder
3. Ability to provide informed consent
4. Age 18 or over
5. Selected for participation based on investigator discretion

Exclusion Criteria:

1. Unable to follow instructions
2. Exhibit significant behavioral problems or impaired cognitive ability
3. Inability to provide consent
4. Non-English speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Theis, MS, OT/L, Principal Investigator — Allina Health System
Locations (1):
- Allina Health Courage Kenny Rehabilitation Institute, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- User Focus Group Participants: Human subjects with spinal cord injury at levels C3 to C5, and ASIA Impairment Scale (AIS) A, B, or C.
  Active Powered Prosthesis (APEX) for Spinal Cord Injury: The Active Powered Prosthesis (APEX) is a proof-of-concept shoulder-elbow-wrist device intended to provide non-invasive active powered robotic assistive movement to upper extremities. Focus group participants will control the APEX device on a test manikin and provide feedback on the device design and function.
Period: Overall Study
Arm/Group | User Focus Group Participants
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | User Focus Group Participants
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: User Ability to Operate the APEX Device
Description: Users evaluate the usability and performance of the APEX device in completion of Activities of Daily Living (ADLs).
Time Frame: Two hours of in-clinic prototype evaluation
Population: Active Powered Prosthesis (APEX) for Spinal Cord Injury: The Active Powered Prosthesis (APEX) is a proof-of-concept shoulder-elbow-wrist device intended to provide non-invasive active powered robotic assistive movement to upper extremities. Focus group participants will control the APEX device on a test manikin and provide feedback on the device design and function. Functions assessed include ability to use voice control features and controlling device to mimic performance of ADLs.
Measure: Count of Participants; unit: Participants
Arm/Group | User Focus Group Participants
Number analyzed (Participants) | 4
Participants
  Change Device Modes using Voice Control | 4
  Control Device to Mimic ADL Performance on Manikin | 4

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | User Focus Group Participants
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT03696927/Prot_SAP_000.pdf